CLINICAL TRIAL: NCT02598908
Title: Collection of Blood Samples for Use in an External Quality Assurance (EQA) Scheme for Thiopurine S-methyl Transferase (TPMT) Activity and Thiopurine Metabolites, 6-thioguanine Nucleotides (6TGN) and 6-methyl Mercaptopurine Nucleotides (6MMPN).
Brief Title: An EQA Scheme for TPMT Activity and Thiopurine Metabolites
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sandwell & West Birmingham Hospitals NHS Trust (Other)
Collaborators: Birmingham Quality (Other)
Responsible Party: Principal Investigator, Jenna Waldron, Principal Clinical Scientist, Sandwell & West Birmingham Hospitals NHS Trust
Other Study IDs: IRAS 194310
Record Dates: First submitted 2015-11-05; First posted 2015-11-06 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: External Quality Control; Thiopurine S-methyl Transferase (TPMT)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Up to 60 mL of EDTA blood will be collected from each of the selected volunteers by trained phlebotomy staff at Sandwell or City hospitals and virology tested just prior to the sample distribution.
  Surplus blood from routine specimens analysed for 6TGN and 6MMPN will be selected on the basis of thiopurine metabolite concentrations of interest and volume of blood remaining.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- NHS staff volunteer donors: Interested staff working within the Pathology Department at SWBH NHS Trust will be provided with written information regarding the proposed EQA scheme and the sample collection procedure. A consent form will be given to staff members, who will be asked to return the signed form within 1 week if they wish to participate. Each participating staff member will be assigned a unique patient identifier to allow for sample results to be anonymised.
  Interventions: Diagnostic Test: Quality control - enzyme activity
- SWBH outpatient donors: A list of SWBH NHS Trust patient TPMT results will be gathered from the Pathology computer system (Telepath). Those with a TPMT activity of interest, measured in the past five years, will be contacted with the agreement of their hospital consultant. Information and consent forms will be sent to the patient either through the post or via their hospital consultant. Each participating patient will be assigned a unique patient identifier to allow for sample results to be anonymised.
  Interventions: Diagnostic Test: Quality control - enzyme activity

INTERVENTIONS:
Diagnostic Test: Quality control - enzyme activity — A blood sample will be collected from patients and staff donors, no more than twice per year.

SUMMARY:
Participation in EQA schemes, where available, is mandatory for the United Kingdom Accreditation Service (UKAS). No EQA scheme currently exists for TPMT and thiopurine metabolites, which is a potential shortcoming of these tests. A pilot of this project has been awarded funding by Clinical Pathology Accreditation (CPA).

The purpose of this work is to collect samples for an EQA scheme for whole blood TPMT (activity and genotype) and thiopurine metabolites, which will be run in collaboration with UK NEQAS (United Kingdom National External Quality Assessment Service), and facilitate a comprehensive world-wide service that enables laboratories providing these tests to fulfil quality goals and ultimately provide optimal patient care.

DETAILED DESCRIPTION:
The thiopurine S-methyl transferase (TPMT) enzyme is involved in the breakdown of thiopurine drugs (such as azathioprine), which are commonly used to treat inflammatory bowel disease and autoimmune diseases. Different individuals in the population have different, genetically determined, levels of TPMT. An individual with absent TPMT activity has a high risk of serious side effects from thiopurine drug treatment. In routine practice, TPMT activity in the blood is measured before starting patients on thiopurine drugs to determine an effective and safe starting dose.

Thiopurine metabolites are the breakdown products of thiopurine drugs and are monitored in the blood of patients on thiopurine drugs to optimise their drug dose.

These tests are performed by laboratories across Britain and around the world. It is important for patient care that the results are of high quality and consistent across different centres. One way of assessing this is through an EQA scheme. No EQA scheme currently exists for TPMT/thiopurine metabolites, which is a potential shortcoming of the tests.

Venous blood collected from NHS staff volunteers and SWBH outpatients, who have had TPMT measured as part of their routine care, will be distributed to participating laboratories every two months. Where it is not possible to find suitable blood donors, pooled surplus blood samples from the laboratory will be used instead. The laboratories will test the samples and return results to UK NEQAS for comparison. A report will be compiled allowing them to compare themselves with other centres and make changes where necessary.

ELIGIBILITY:
Inclusion Criteria:

* Pathology staff member - able to donate 60 mL of venous blood.
* SWBH NHS Trust outpatients - have had TPMT activity measured within last 5 years. Consultant happy for them to be contacted. Able to consent and donate 60 mL of blood.

No known Hep B or C, HIV, syphilis or cytomegalovirus infection.

Exclusion Criteria:

* Donors for each distribution will be under no obligation to participate if they are no longer willing to. Only volunteers able to give informed consent themselves will be recruited (i.e. no children or adults lacking the capacity to consent themselves).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Interested staff working within the Pathology Department at SWBH NHS Trust
  A list of SWBH NHS Trust patient TPMT results will be gathered from the Pathology computer system. Those with a TPMT activity of interest, measured in the past five years, will be contacted with the agreement of their hospital consultant.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-02-24 (Actual); Primary Completion 2022-02-24 (Estimated); Study Completion 2022-02-24 (Estimated)

PRIMARY OUTCOMES:
TPMT activity | 5 years EQA scheme
  TPMT activity will be determined by participating laboratories

SECONDARY OUTCOMES:
Thiopurine metabolites | 5 years EQA scheme
  Thiopurine metabolites will be determined by participating laboratories

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Berg, FRCPath, MBA, Study Director — SWBH, Pathology director
Locations (1):
- Department of Biochemistry, City Hospital, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Not applicable. Results will be analysed anonymised.

REFERENCES:
- See also: Birmingham quality UK NEQAS — http://www.birminghamquality.org.uk/
- See also: SWBH Pathology laboratory — http://www.cityassays.org.uk/